CLINICAL TRIAL: NCT05404490
Title: Efficacy of Bupivacain Local Infiltration for the Management of Pain During Cesarean Section. Randomized, Single Blind, Controlled Trial
Brief Title: Efficacy of Bupivacain Local Infiltration for the Management of Pain During Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Chair of the Research Department, Saint Thomas Hospital, Panama
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-575
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Pain, Postoperative
Keywords: Cesarean section; Postoperative Pain; Bupivacain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupivacaine (Experimental): 20 mL of bupivacaine 0.5% will be infiltrated. 10 mL will be infiltrated in the inferior border and 10 mL in the superior border of the subcutaneous cellular tissue.
  Interventions: Drug: Bupivacain
- Placebo (Placebo Comparator): 20 mL of Normal Saline Solution will be infiltrated. 10 mL will be infiltrated in the inferior border and 10 mL in the superior border of the subcutaneous cellular tissue.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bupivacain — 20 mL of bupivacaine 0.5% will be infiltrated. 10 mL will be infiltrated in the inferior border and 10 mL in the superior border of the subcutaneous cellular tissue.
  Arms: Bupivacaine
Drug: Placebo — 20 mL of Normal Saline Solution will be infiltrated. 10 mL will be infiltrated in the inferior border and 10 mL in the superior border of the subcutaneous cellular tissue.
  Arms: Placebo

SUMMARY:
This study aims to evaluate the effect of local administration of bupivacain in the cesarean section incision for postoperative pain control, using the visual analogue pain scale (VAS) and assessing the need for rescue analgesia after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≥ 36 weeks
* Elective cesarean section
* Transverse segmental caesarean section Pfannenstiel type
* Spinal anesthesia
* Maternal age 18 to 45 years
* Any gravaparity
* Patient ASA I or II

Exclusion Criteria:

* Any patient who does not meet the inclusion criteria.
* Emergency cesarean section
* History of chronic or neuropathic pain
* Patient with cardiopulmonary disease
* Known allergies to the drugs used in the study
* Patient who does not wish to participate in the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Post operative pain | 72 hours
  Level of pain described using a Visual Analogue Scale (VAS) Lower value: 0 (no pain) Higher value: 10 (worst pain possible)

SECONDARY OUTCOMES:
Need for rescue medication | 72 hours
  Number of participants that required an additional analgesic for pain control

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Thomas H, Panama City, Provincia de Panamá, Panama

IPD SHARING:
Plan to Share IPD: No